CLINICAL TRIAL: NCT04415242
Title: IMPACT OF OPERATIVE POSITIONING ON THE DEVELOPMENT OF SHOULDER PAIN AFTER PULMONARY LOBECTOMY BY VATS
Acronym: POVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Geraud Galvaing, MD, MSc, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-3430, 21919
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Post-thoracotomy Pain Syndrome
Keywords: VATS; shoulder pain; pulmonary resection
MeSH Terms: conditions — Shoulder Pain | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suspension group (Active Comparator): Arm on the side operated at 90 ° abduction, 90 ° anti-drive, resting on an arm support.
  Interventions: Other: positioning
- supported group (Experimental): Arm on the operated side at 0 ° abduction, 90 ° anti-pulsation, resting on an adjustable support arm support located opposite the patient's head.
  Interventions: Other: positioning

INTERVENTIONS:
Other: positioning — different positioning prior surgery

SUMMARY:
The investigators want to be able to show a 66% decrease in the incidence of shoulder pain in the "support" group compared to the "suspension" group.

DETAILED DESCRIPTION:
The position currently used in cases of pulmonary lobectomies by videothoracoscopy is an extension associated with an abduction of the shoulder on the side operated by suspension of the thoracic limb in a trampoline-type arm support with an angulation of more than 90 ° of the shoulder in the saggital and frontal planes.

The investigators wish to prospectively and randomly compare this position currently used in the thoracic surgery service of the IUCPQ with a 2nd position which seems less restrictive for all the joints of the shoulder joint complex in which the patient's arm rests on a support placed in front of the patient's face. It follows from this position of the joint degrees less than or equal to 90 ° in all planes. This new position is not experimental, but not normally used in thoracic surgery at the IUCPQ.

ELIGIBILITY:
Inclusion Criteria:

* Any patient in whom the management of a bronchopulmonary cancer, or his strong suspicion, justifies a bilobectomy, a lobectomy or a segmentectomy by videothoracoscopy.

Exclusion Criteria:

* surgery extended to the chest wall, including extra-pleural resections,

  * Pleurectomy,
  * Chronic pain patient suffering from chronic pain preoperatively,
  * Fibromyalgia patient,
  * Chronic taking of analgesic or anti-inflammatory medications during the preoperative period, namely taking at least daily for more than 4 weeks,
  * Patient with a history of orthopedic surgery of the upper limb ipsilateral to the surgery,
  * Patient with mechanical limitation of the joint range of the upper limb ipsilateral to surgery,
  * Non-French speaking patient,
  * Pregnant woman,
  * Patient under 18-year-old,
  * Patient whose BMI is greater than or equal to 35 kg / m2
  * Glomerular filtration rate less than <50 ml / min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
post thoracoscopy shoulder pain measured on the Visual Pain Scale | from the recovery unit to post-operative day 2
  postoperative shoulder pain measured on the Visual Pain Scale, its precise location on the patient's body will also be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Barak M, Ziser A, Katz Y. Thoracic epidural local anesthetics are ineffective in alleviating post-thoracotomy ipsilateral shoulder pain. J Cardiothorac Vasc Anesth. 2004 Aug;18(4):458-60. doi: 10.1053/j.jvca.2004.05.025. PMID 15365928